CLINICAL TRIAL: NCT06728007
Title: Nephrological Outcome and Associated Congenital Anomalies in Pediatric Patients with Horseshoe Kidney
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HSK-PED-23-01
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Horseshoe Kidney
Keywords: Horseshoe Kidney; Congenital anomalies; Children; CAKUT
MeSH Terms: conditions — Fused Kidney; Congenital Abnormalities; Cakut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A retrospective, observational multicentre trial on the nephrological outcome and associated congenital anomalies in children with Horseshoe Kidney.

DETAILED DESCRIPTION:
Congenital abnormalities of the kidney and urinary tract (CAKUT) represent the main cause of CKD in children. Among them, the horseshoe kidney (HSK) represents one of the most frequent and is characterised by the presence of two distinct, functioning kidneys positioned on each side of the spine, fused together at one of the poles. The incidence of this condition is approximately 1 case every 400-600 new births with a prevalence in the male sex with a ratio of 2:1. Even though these children aregenerally asymptomatic and the diagnosis is often incidental , some may develop symptoms due to complications, such as infections, nephrolithiasis and urinary tract obstruction. More rarely risks of neoplastic degeneration and renal damage are described following trauma to the abdomen and lumbosacral spine. This condition is also associated in up to a third of cases with other abnormalities: the most frequent affect the urinary tract and genitals; however, abnormalities affecting other organs or systems as well as well-defined syndromic pictures. Due to its frequent asymptomatic nature, horseshoe kidney is historically considered a condition with a good prognosis and rarely as a risk factor capable of reducing survival or predisposing the kidney to long-term damage.

The primary objective of the study is:

To assess the 'nephrological outcome' understood as 'prevalence of patients who developed' and 'survival time free from": chronic renal failure, proteinuria, hypertension nephrolithiasis, UTI, renal neoplasms and renal trauma.

The secondary objectives of the study are:

1. Prevalence of congenital and associated genito-urinary and systemic abnormalities;
2. Description of renal anatomical features;
3. Assessment of the usefulness of second level radiological investigations (VCUG, static renal scintigraphy, ddynamic renal scintigraphy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed ultrasound and/or scintigraphic diagnosis of horseshoe kidney;
* Patients with an age at first assessment of between 0 and 18 years;
* Obtaining written Informed consent.

Exclusion Criteria:

* Patients with a definitive diagnosis of another form of CAKUT during the diagnostic pathway.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients followed at the participating centres from 01/01/2012 to 31/12/2021 for a nephro-urological pathology will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Chronic kidney disease | at baseline
  Defined as a reduction in eGFR <90ml/min/1.73m2, calculated using the Schwartz formula(18) corrected for age:
  * δ= 0.45 for children <1 yr
  * δ= 0.55 for children of both sexes from 2 to 12 yrs and for female children aged 13 to 18 yrs
  * δ= 0.70 for children aged 13 to 18 yrs
  The different stages of chronic kidney have been further defined according to eGFR:
  * Stage I: >90ml/min/1.73m2
  * Stage II: between 89 and 60ml/min/1.73m2
  * Stage III: between 59 and 30ml/min/1.73m2
  * Stage IV: between 30 and 15ml/min/1.73m2
  * Stadio V: lower than15ml/min/1.73m2 or patient in dialysis
Proteinuria | at baseline
  Defined as the urinary protein:creatinine ratio (mg/mg) >0.5 in chilrden up to 2 yrs of age and >0.2 in chilrden older than 2 yrs
Hypertension | at baseline
  Arterial blood pressure ≥95th percentile for sex, age and height, on at least three different readings

SECONDARY OUTCOMES:
Urinary tract infections | at baseline
  Confirmed by urine analysis and urine culture in a compatible clinical picture
Nephrolithiasis | at baseline
  Documented finding by imaging techniques (ultrasound and/or CT) of formations compatible with lithiasis formation
Renal neoplasms | at baseline
  Diagnosis confirmed by imaging and histology of the neoplasm of renal origin (especially Wilms' tumour)
Renal anatomical features | at baseline
  Renal length measured as bipolar diameter with renal hypoplasia defined as the presence of kidneys with DBP <5° centile reference for age and height
Renal anatomical features | at baseline
  Ultrasound description of abnormalities of the renal parenchyma with renal dysplasia defined by the presence of alterations such as: hyperechogenicity, reduced cortico-middular differentiation, reduced cortical thickness due to age, presence of multiple cystic formations
Renal trauma | at baseline
  Presence of instrumentally documented renal lesions (ultrasound and/or CT scan) following a traumatic episode

CONTACTS AND LOCATIONS:
Overall Officials: Claudio La Scola, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy